CLINICAL TRIAL: NCT07303400
Title: Assessment of the Effectiveness of a Prototype Diagnostic System of Bacterial Respiratory Infections Based on Real-time Sequencing
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Stefano Gaiarsa, Researcher, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: ASAP
Record Dates: First submitted 2025-12-02; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-08

CONDITIONS: Lower Resp Tract Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The objective of this project is to test the efficiency of a novel developed protocol for direct real-time metagenomic sequencing of Lower Respiratory Infection samples. The investigators aim to assess the anticipation time, compared to the traditional culturing methods and the accuracy, compared to gold standards

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to provide written informed consent prior to performing the study procedures
2. Patients older than 18 years of age
3. Suspected bacterial Lower Respiratory Infection (LRI)
4. 500µL of lower respiratory tract sample (e.g. Bronchoalveolar lavage) are available after the routine diagnostic procedures are over

Exclusion Criteria:

1. Low amount of leftover specimen
2. Complex diagnosis: clinicians could require further analysis after the first diagnosis is produced
3. A sample of the same patient has been already included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients tested for Lower Respiratory tract infections using bronchoalveolar lavage samples
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
test positivity | Baseline
  assess the effectiveness in detection of positive (Gram+ vs Gram- vs mixed culture samples) vs negative samples
species identification | Baseline
  Assess the effectiveness in recognizing the correct bacterial species

SECONDARY OUTCOMES:
anticipation time | Baseline
  Measure the anticipation time of the novel protocol vs gold standard (culturing)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy